CLINICAL TRIAL: NCT01780701
Title: Imaging Prostatic Lipids to Distinguish Aggressive Prostate Cancer
Brief Title: Magnetic Resonance Spectroscopic Imaging Study of Prostatic Fats to Distinguish the Difference Between High and Low Risk Prostate Cancer
Acronym: MRSI+RRP
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Portland VA Medical Center (U.S. Federal Agency); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jackie Shannon, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: IRB00008458; W81XWH-12-1-0168 (Other Grant/Funding Number: Dept of Defense); 2978 (Other: Portland VA Medical Center IRB); 8458 (Other: Oregon Health & Science University IRB); Log #A-17208 (Other: Dept of Defense Human Research Protection Office); PC110361 (Other: Dept of Defense)
Record Dates: First submitted 2013-01-07; First posted 2013-01-31 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer aggressiveness; magnetic resonance imaging; fatty acid synthase
MeSH Terms: conditions — Prostatic Neoplasms; Prostate Cancer, Hereditary, 7 | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Prostatic fluid and Prostatectomy tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk prostate cancer patients: Men who have been recently diagnosed with high risk prostate cancer (Gleason score 7 and above) and who choose prostate removal for their cancer treatment will undergo Magnetic Resonance Spectroscopy Imaging (MRSI) with rectal probe at the Oregon Health & Science University's Advanced Imaging Research Center.
  Interventions: Procedure: Magnetic Resonance Spectroscopy Imaging with rectal probe
- Low risk prostate cancer patients: Men who have been recently diagnosed with low risk prostate cancer (Gleason score 7 [3+4] and below) and who choose prostate removal for their cancer treatment will undergo Magnetic Resonance Spectroscopy Imaging (MRSI) with rectal probe at the Oregon Health & Science University's Advanced Imaging Research Center.
  Interventions: Procedure: Magnetic Resonance Spectroscopy Imaging with rectal probe

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopy Imaging with rectal probe
  Other Names: Magnetic Resonance Spectroscopy Imaging; MRSI; Magnetic Resonance Imaging; MRI

SUMMARY:
A prostate cancer diagnosis starts a list of events that often leads to fast-moving treatment, thought by many to result in vast over-treatment of this disease. So, discovery of different diagnostic methods that allow clinicians to identify slow-growing from potentially fast-growing disease prior to or at the time of prostate biopsy could result in early and suitable treatment for men at greatest risk, while greatly decreasing the number of biopsies, surgical procedures, hormonal and chemotherapeutic treatments, cost, and patient worry, for those with more slow-growing disease.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer diagnosis prior to treatment
* Age 21 years or older
* Signed informed subject consent
* Prostatectomy as planned prostate cancer treatment

Exclusion Criteria:

* Men who do not choose prostatectomy
* Men who have undergone any neoadjuvant therapy
* Men who have cardiac pacemakers or other implanted electronic devices
* Men who have any surgically implanted metal
* Men who have had any surgical procedure that precludes placement of endorectal probe
* Indication of dementia or memory issues listed on problem list
* Men who indicate exposure to ocular metal fragments; confirmed by positive ocular x-ray
* Men who are taking newly-prescribed (within 6 months of enrollment) lipid control medications

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all men newly-diagnosed with prostate cancer at the Portland VA and OHSU Urology clinics
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with increased intraprostatic lipid concentration | Up to 3 years
  Determine the correlation between the amount of intraprostatic lipid using 1H (proton) magnetic resonance spectroscopic imaging (MRSI) with an endorectal coil obtained prior to prostatectomy with fatty acid synthase protein expression measured in benign and cancer tissue from prostatectomy samples.

SECONDARY OUTCOMES:
Number of participants with increased tumor aggressiveness | Up to 3 years
  Identify the association between fatty acid synthase protein expression in prostatectomy samples, intraprostatic lipid as measured by 1H MRSI, and prostate tumor aggressiveness.

OTHER OUTCOMES:
Number of participants with accumulation of lipid intermediates and proteins | Up to 3 years
  To quantify the association between key metabolic intermediates involved in lipid metabolism, mitochondrial function, inflammation, and apoptosis in prostatectomy samples and fatty acid synthase protein expression, intraprostatic lipid and tumor aggressiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — Oregon Health and Science University; Jonathan Q Purnell, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Portland VA Medical Center, Portland, Oregon
  - Oregon Health & Science University Advanced Imaging Research Center, Portland, Oregon